CLINICAL TRIAL: NCT00281463
Title: Impact of Pushrim Activated Power Assist Wheelchairs on Mobility Among People With Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rory Cooper, Director; Pittsburgh VA Rehabilitation Research & Development Center, VA Pittsburgh Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 01103, 010842; H133N000019
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Wheelchair Users
Keywords: wheelchair; spinal cord injury; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pushrim Activated Power Assist Wheelchair (Experimental): Participants will be asked to propel both their own chair and a pushrim activated power assist wheelchair on a computer controlled wheelchair dynamometer.
  Interventions: Device: Pushrim Activated Power Assist

INTERVENTIONS:
Device: Pushrim Activated Power Assist — The PAPAW is an electrically-powered add-on unit for common manual wheelchairs. The unit automatically supplements the users manual pushrim input with additional rear-wheel torque for up to six kilometers/hour traveling velocity. The amount of added torque is provided proportional to the user input to the pushrims. Movement and braking assistance is provided for both forward and rearward travel. Several types and sizes are available based on users operating strength, needs and anthropometry. The PAPAWs to be tested during this study will be the JWII (Yamaha Motor Corporation).

SUMMARY:
The purpose of this three phase study is to evaluate a Pushrim Activated Power Assist Wheelchair (PAPAW). Phase I will examine whether the steady-state, metabolic energy efficiency for propelling a manual wheelchair with and without the device will be significantly different. In Phase II, wheelchair users will evaluate the PAPAW over activities of daily living course to determine its usability and acceptability and to identify areas for future development. Finally, in phase III, comparison of activities of daily living in the community will be made between the subjects when using their personal wheelchair and a PAPAW.

DETAILED DESCRIPTION:
Objectives:

The purpose of this three phase study is to evaluate a Pushrim Activated Power Assist Wheelchair (PAPAW). Phase I will examine whether the steady-state, metabolic energy efficiency for propelling a manual wheelchair with and without the device will be significantly different. In Phase II, wheelchair users will evaluate the PAPAW over activities of daily living course to determine its usability and acceptability and to identify areas for future development. Finally, in phase III, comparison of activities of daily living in the community will be made between the subjects when using their personal wheelchair and a PAPAW.

Research Design:

This is a repeated measures design type study, conducted in different locations for each phase: a biomechanics laboratory, an ADL driving course, and the participants' home environment. Analyzed variables include: metabolic energy expenditures, stroke frequency, upper extremity joint range of motion, participant responses to a visual analog survey, average speed, and actual daily driving time spent in either wheelchair, and daily distance traveled. Subjects will act as their own controls.

Methodology:

Full-time wheelchair users with tetraplegia between the ages of 18 and 65 will be recruited for the study. They will be free of pressure sores, free from any shoulder pain that would prevent them from propelling a manual wheelchair, and have no history of cardiopulmonary disease. A maximum of 50 subjects (fifteen for Phase I and II, and 15 or Phase III, and five for subject drop-out) will be recruited. In Phase I, participants will be asked to propel a PAPAW and their own wheelchair, attached to a wheelchair roller system through three resistance conditions. In Phase II, participants will be asked to propel both wheelchairs over activities of daily living. Finally, Phase III consists of a four-week trial including a two-week test with subjects' own wheelchairs (i.e. own chair trial) and a two-week test where they were provided with the PAPAW (i.e. PAPAW trial). The order of the own chair trial and the PAPAW trial will be randomized.

Clinical Relationship:

For individuals with tetraplegia, PAPAWs reduce energy demands, stroke frequency, and overall joint range of motion when compared to traditional manual wheelchair propulsion. In addition, PAPAWs have the potential to improve the functional capabilities during certain activities of daily living as well as community participation of individuals with tetraplegia. Use of this device could help maintain overall physical capacity while reducing the risk for pain and injuries to the upper extremities.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 65 years of age
* Full time wheelchair user
* Diagnosis of Tetraplegia

Exclusion Criteria:

* Pressure sores
* Shoulder pain that would prevent them from propelling a manual wheelchair
* History of cardiopulmonary disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2001-11; Primary Completion 2007-03 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rory A Cooper, PhD, Principal Investigator — Human Engineering Research Laboratories
Locations (1):
- Human Engineering Research Laboratories, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pushrim Activated Power Assist Wheelchair
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pushrim Activated Power Assist Wheelchair
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Consumption
Time Frame: in-lab visit when propelling on a computer controlled wheelchair dynamometer
Population: personal w/c (.9 m/s, 10 W)
Measure: Mean (Standard Deviation); unit: VO2 (ml/min)
Groups:
- Pushrim Activated Power Assist Wheelchair: Participants were asked to propel both their own chair and a pushrim activated power assist wheelchair on a computer controlled wheelchair dynamometer.
Arm/Group | Pushrim Activated Power Assist Wheelchair
Number analyzed (Participants) | 15
VO2 (ml/min) | 625 (316)

2. Primary Outcome: Oxygen Consumption
Time Frame: in-lab visit when propelling on a computer controlled wheelchair dynamometer
Population: PAPAW (.9 m/s, 10 W)
Measure: Mean (Standard Deviation); unit: VO2 (ml/min)
Arm/Group | Pushrim Activated Power Assist Wheelchair
Number analyzed (Participants) | 15
VO2 (ml/min) | 415 (204)

ADVERSE EVENTS:
Arm/Group | Pushrim Activated Power Assist Wheelchair
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No